CLINICAL TRIAL: NCT03795194
Title: A Prospective, Randomized Trial of Antibiotic Duration in Post-appendectomy Abscess
Brief Title: Antibiotic Duration in Post-appendectomy Abscess
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to low enrollment.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-055
Record Dates: First submitted 2018-07-19; First posted 2019-01-07 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Complicated Appendicitis; Perforated Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ampicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 8-day (Other): 8-day course of ampicillin clavulanate antibiotic
  Interventions: Drug: ampicillin/clavulanate
- 4-day (Other): 4--day course of ampicillin clavulanate antibiotic
  Interventions: Drug: ampicillin/clavulanate

INTERVENTIONS:
Drug: ampicillin/clavulanate — FDA-approved antibiotic
  Other Names: Augmentin

SUMMARY:
This is a randomized study of patients 2-17 years old who are diagnosed with perforated appendicitis and develop an abscess after laparoscopy that is subsequently drained. Patients will be randomized to either receive an 8-day or a 4-day course of antibiotics. The aim of this study is to determine whether duration of antibiotic treatment at discharge demonstrates significant differences in clinical outcomes.

DETAILED DESCRIPTION:
The central aim of this study is to determine whether duration of antibiotic treatment at discharge demonstrates significant differences in primary and secondary clinical outcomes. Specifically, this research aims to determine whether the readmission rate and length of stay for pediatric patients diagnosed with perforated appendicitis who form a post-laparoscopic abscess that is treated with percutaneous drainage and are treated with a 8-day oral antibiotic regimen at discharge is significantly different from those treated with a fixed 4-day regimen at discharge.

This study includes patients ages 2-17 years old who present with perforated appendicitis-as diagnosed at laparoscopy and photographed as either a hole or as feces in the abdomen-and who develop an abscess after laparoscopy that is treated with percutaneous drainage.

All post-laparoscopic abscess patients will receive the standard of care for antibiotic therapy at Phoenix Children's Hospital-IV ceftriaxone/metronidazole-until afebrile and tolerating food. All patients will be treated with the PCH standard of care and receive in-patient treatment for abscess until afebrile.

At discharge, study patients will be randomly assigned to either an 8-day ampicillin/clavulanate regimen or a 4-day ampicillin/clavulanate regimen. Pediatric patients who are allergic to ampicillin will be excluded from the study. Patients will be followed thirty days post discharge to assess clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 to 17 years of age
* Diagnosis of perforated appendicitis at laparoscopy
* Development of a post-appendectomy abscess that is treated with percutaneous drainage.

Exclusion Criteria:

* Patients who are allergic to ampicillin

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Egan, MD, Principal Investigator — Phoenix Children's
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 8-day | 4-day
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (8-day); Arm B (4-day): In this study, all patients will be treated with the hospital standard of care and receive in-patient treatment for abscess until afebrile and tolerating food for 24 hours. After percutaneous drainage of the abscess, the patient will be randomly assigned to receive either an 8-day regimen (arm A) or a 4-day regimen (arm B) of antibiotics (Diagram 1). Patients will remain on IV ceftriaxone/metronidazole or other broad spectrum antibiotic equivalent until afebrile and tolerating food for 24 hours. Patients will complete their assigned 4- or 8-day regimen with oral ampicillin clavulanate or other broad spectrum antibiotic equivalent. If patients are not afebrile at the completion of their assigned regimen, prescribing an extended course of antibiotics is at the discretion of the treating surgeon. A prescribed oral course of antibiotics may be finished in the hospital or at home if patient is discharged.
- Total: Total of all reporting groups
Arm/Group | Arm A (8-day) | Arm B (4-day) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.34 (2.48) | 9.65 (3.56) | 12.09 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmission Rate
Description: Rate of readmission to the hospital after abscess drainage.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (8-Day) 30-day Readmission Rate: Rate of readmission to hospital following source control of abscess when treated with antibiotics for 8 days.
- Arm B (4-Day) 30-day Readmission Rate: Rate of readmission to hospital following scource control of abscess when treated with antibiotics for 4 days.
Arm/Group | Arm A (8-Day) 30-day Readmission Rate | Arm B (4-Day) 30-day Readmission Rate
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

2. Primary Outcome: Length of Hospital Stay
Description: How many days patient stays in the hospital if and when they are readmitted after their abscess drainage.
Time Frame: 30 days
Population: Participants were not readmitted to the hospital after abscess drainage.
Groups:
- Arm A (8-day): Arm A hospital length of stay if readmitted following abscess drainage.
- Arm B (4-day): Arm B hospital length of stay if readmitted following abscess drainage.
Arm/Group | Arm A (8-day) | Arm B (4-day)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed 30 days post-discharge after abscess drainage.
Arm/Group | 8-day | 4-day
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
Low enrollment. Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT03795194/Prot_SAP_000.pdf